CLINICAL TRIAL: NCT02952794
Title: Endoscopic Submucosal Dissection (ESD) and Endoscopic Mucosal Band Ligation (EMBL) for Early Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Professor, Fudan University
Other Study IDs: S2015101
Record Dates: First submitted 2015-06-22; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Early Cancer
Keywords: endoscopic submucosal dissection (ESD); endoscopic mucosal band ligation (EMBL)
MeSH Terms: conditions — Neoplasms | interventions — Endoscopic Mucosal Resection; s-formylglutathione hydrolase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ESD: endoscopic submucosal dissection (ESD)for early cancer
  Interventions: Procedure: endoscopic submucosal dissection (ESD) and endoscopic mucosal band ligation (EMBL) for early cancer
- EMBL: endoscopic mucosal band ligation (EMBL) for early cancer
  Interventions: Procedure: endoscopic submucosal dissection (ESD) and endoscopic mucosal band ligation (EMBL) for early cancer

INTERVENTIONS:
Procedure: endoscopic submucosal dissection (ESD) and endoscopic mucosal band ligation (EMBL) for early cancer

SUMMARY:
To compare the treatment methods of endoscopic submucosal dissection (ESD) and endoscopic mucosal band ligation (EMBL) for early cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early neoplasm in the gastrointestinal tract

Exclusion Criteria:

* Patients who can not meet the surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: endoscopic submucosal dissection (ESD) and endoscopic mucosal band ligation (EMBL) for early cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Center, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China